CLINICAL TRIAL: NCT02263066
Title: Retrospective Study in Chinese Pediatric Hemophilia A Patients With rFⅧ Contained Regular Prophylaxis
Acronym: ReCARE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17653
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Chinese hemophilia A pediatric patients with medical records who had accepted regular prophylaxis, totally/partially with rFⅧ between Nov. 1st 2007 and May 31st 2013
  Interventions: Biological: BAY14-2222_Kogenate-FS FVIII

INTERVENTIONS:
Biological: BAY14-2222_Kogenate-FS FVIII — Depends on Doctor's decision

SUMMARY:
To assess and describe real-life treatment choices for rFⅧ contained regular prophylaxis/bleeding prevention treatment in pediatric hemophilia patients in China (2007-2013)

ELIGIBILITY:
Inclusion Criteria:

* Male, 2-<18 years Hemophilia A, based on documented prior testing and/or screening laboratory Patients who had received regular prophylaxis/bleeding prevention treatment, totally/partially with rFⅧ. Regular prophylaxis/bleeding prevention treatment is defined as that proportion of weeks (≥2 infusion/week) of total treatment weeks≥80%[10] , and total duration ≥12 weeks. During the regular prophylaxis period, if there were consecutive 4 weeks that <2 infusion/week, the beginning day of the 4 weeks is defined as the end of regular prophylaxis.

Available patient medical data record Written informed consent by parent/legal representative. Consent should be sought from subjects if appropriate

Exclusion Criteria:

* Patients with measurable inhibitor activity at baseline and history of FVIII inhibitor antibody formation (≥0.6BU by Bethesda assay at two different time points, documentation must be available) Any individuals with another bleeding disease that is different from hemophilia A (e.g, von Willebrand disease, hemophilia B)

Ages: 2 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: About 300 at most hemophilia boys (2-<18 years) in the representative hemophilia treatment centers (HTCs) with available medical data record, having received rFVIII contained regular prophylaxis between Nov. 1st 2007 and May 31st 2013 will be enrolled from about 15 centers.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Duration of regular prophylaxis | Up to 1.5 years
Prophylaxis infusion dose | Up to 1.5 years
Percentage of rFVIII usage in prophylaxis | Up to 1.5 years

SECONDARY OUTCOMES:
Bleeding frequency | Up to 1.5 years
Joint radiographic score | Up to 1.5 years
Joint physical examination score | Up to 1.5 years
Quality of life by questionnaire | Up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China

REFERENCES:
- [Derived] Li C, Zhang X, Zhao Y, Wu R, Hu Q, Xu V, Sun J, Yang R, Li X, Zhou R, Lian S, Gu J, Wu J, Hou Q. Status and trend analysis of prophylactic usage of recombinant factor VIII in Chinese pediatric patients with hemophilia A: ReCare - a retrospective, phase IV, non-interventional study. Curr Med Res Opin. 2017 Sep;33(9):1571-1578. doi: 10.1080/03007995.2017.1333489. Epub 2017 Jun 21. PMID 28532239
- [Derived] Li C, Zhang X, Zhao Y, Wu R, Hu Q, Xu W, Sun J, Yang R, Li X, Zhou R, Lian S, Gu J, Wu J, Hou Q. Long-term efficacy and safety of prophylaxis with recombinant factor VIII in Chinese pediatric patients with hemophilia A: a multi-center, retrospective, non-interventional, phase IV (ReCARE) study. Curr Med Res Opin. 2017 Jul;33(7):1223-1230. doi: 10.1080/03007995.2017.1310720. Epub 2017 Apr 25. PMID 28326849